CLINICAL TRIAL: NCT07188662
Title: Role of Multimodal Prehabilitation Program in Improving Surgical Outcomes for Women Undergoing Gynecologic Oncology Surgery
Brief Title: Multimodal Prehabilitation Program for Women Undergoing Gynecologic Oncology Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya M. Abdelhafez, lecturer of maternity, gynecological and obstetric nursing, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMPPGOS
Record Dates: First submitted 2025-07-11; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Gynecologic Oncology Patient
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (No Intervention): Conventional group (woman received hospital care at previous year as a retrospective sample to prevent risk of bias) equal 70 woman
- Prehabilitation group (Experimental): Prehabilitation group (woman who will receive prehabilitation care combine with ERAS post-operative care as a prospective sample) equal 70 woman
  Interventions: Procedure: group (B) Prehabilitation care combine with ERAS post-operative care

INTERVENTIONS:
Procedure: group (B) Prehabilitation care combine with ERAS post-operative care — intervention will includes receiving prehabilitation care combine with ERAS post-operative care.
  Arms: Prehabilitation group

SUMMARY:
The goal of this clinical trial is to evaluate the role of multimodal Prehabilitation program on improve surgical outcomes after gynecological oncology surgery.

DETAILED DESCRIPTION:
Multimodal prehabilitation program focused on improving woman physical and psychological wellbeing before gynecological oncology surgery. Multimodal prehabilitation refers to a combination of preoperative interventions targeting physical, nutritional, psychological, and medical optimization. This program included various element such preoperative physical exercise, nutritional support, psychological counselling, social support and education about surgical processes. Multimodal Prehabilitation programs play an important role in improving surgical outcomes after gynecological oncology surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed woman with gynecologic cancer by imaging &histopathology
* Accept participation in the study.

Exclusion Criteria:

* Patient with advanced and metastatic stage
* Patient who received neoadjuvant chemotherapy
* Patient who have psychological disorder such as suicidal attempt
* Patient who have cerebral stroke, hemiplegia or paralyses

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
changing the postoperative morbidity | "up to 30 days postoperative"
  compare the 30 days postoperative morbidity of the prehabilitation and conventional group, it included (Assess the post-operative complications by using Clavien-Dindo classification; from Grade I-IV; higher grades indicate more severe complications.)
changing the postoperative mortality | "up to 30 days postoperative"
  compare the 30 days postoperative mortality of the prehabilitation group and conventional group.
Pain intensity measured by the Visual Analog Scale (VAS) for pain. | "up to 30 days postoperative"
  compare the 30 days postoperative Pain intensity; Unit of Measure: Units on a scale (0-10 cm).
  Scale: 0 = no pain, 10 = worst pain imaginable; higher scores indicate worse pain of the prehabilitation group and conventional group.

SECONDARY OUTCOMES:
change the length of the hospital stay | up to 5 days post-operative
  compare the days of the hospital stay between the prehabilitation group and conventional group to measure the effect of the intervention program in changing the length of hospital stays (Number of days from surgery until hospital discharge).
Enhance the physical state of gynecological oncology patient using the Eastern Cooperative Oncology Group (ECOG) | through the postoperative period within two hours up-to 30 days after surgery
  - Eastern Cooperative Oncology Group (ECOG) is a performance method used to assess a cancer patient's level of functioning and ability to care for themselves, work, and carry out daily activities. ECOG Performance Status Scale included 5 grades from 0- 5
  * Grade 0: Fully active, able to carry all activities without restriction.
  * Grade 1: Restricted in physically and able to do light work
  * Grade 2: Ambulatory and capable of self-care, but unable to carry out any work activities; up >50% of waking hours.
  * Grade 3: Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  * Grade 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  * Grade 5: Dead.
Enhance the psychological wellbeing of gynecological oncology patient | up-to 15 days preoperatively & up to 30 days post operatively]
  - measure the Psychological aspect by using DASS21(Depression, Anxiety, and Stress Scale - 21 items):
  . 1- Depression
  * Unit of Measure: Units on a scale (0-42).
  * Scale: Higher scores indicate worse depression. 2- Anxiety
  * Unit of Measure: Units on a scale (0-42).
  * Scale: Higher scores indicate worse anxiety. 3- Stress
  * Unit of Measure: Units on a scale (0-42).
  * Scale: Higher scores indicate worse stress
assess and changing the Nutritional Status of the prehabilitation group | up-to 30 days postoperative
  Nutritional Status measured through the following:
  1. Nutritional Status - Height/m Description: Patient height measured in meters.
  2. Nutritional Status - Weight/kg Description: Patient body weight measured in kilograms.
     * weight and height combined to report BMI in kg/m^2
assess and changing the Nutritional Status of the prehabilitation group | up-to 30 days postoperative
  Nutritional Status measured through:
  - Clinical Signs using Patient-Generated Subjective Global Assessment (PG-SGA): The PG-SGA is a subjective nutritional assessment tool used in oncology; include questions about:
  * Weight change (past 1 month and 6 months (increased 0 or decreased 1
  * Eating patterns changed over last weeks or months (normal, less than normal, only liquids, very little, etc.)
  * Gastrointestinal Symptoms affecting intake (e.g., nausea, vomiting ,pain, diarrhea, etc.)
  * Functional capacity& activity (normal activity, reduced, bed/chair bound, etc.) Scoring system of PG-SGA: A)Well-nourished (0-3) B)Moderately malnourished 4-8 C)Severely malnourished more then >9
improve the Cardiopulmonary fitness of gynecological oncology patient after surgery | up-to 15 days preoperatively & up to 30 days post operatively]
  Cardiopulmonary Fitness measured by use of:
  1- 6-Minute Walk Test (6MWT) Distance
  * Description: Distance walked in meters.
  * Time Frame: Up to 30 days post operatively .
improve the Cardiopulmonary fitness of gynecological oncology patient after surgery | up-to 15 days preoperatively & up to 30 days post operatively]
  Cardiopulmonary Fitness measured by use of:
  - VO2max (calculated): Estimated VO2max in mL/kg/min using the predictive equation from 6MWT distance and BMI.
  * Time Frame: up to 30 postoperatively
  * Unit of Measure: mL/kg/min.
improve the Cardiopulmonary fitness of gynecological oncology patient after surgery | up-to 15 days preoperatively & up to 30 days post operatively]
  Cardiopulmonary Fitness measured by use of:
  - Fatigue - Visual Analog Scale (VAS) for Fatigue
  * Time Frame: Up to 15 days preoperatively -operative.
  * Unit of Measure: Units on a scale (0-10 cm).
  * Scale: 0 = no fatigue, 10 = worst fatigue imaginable; higher scores indicate worse fatigue.
improve the Cardiopulmonary fitness of gynecological oncology patient after surgery | up-to 15 days preoperatively & up to 30 days post operatively]
  Cardiopulmonary Fitness measured by use of:
  - Dyspnea - Visual Analog Scale (VAS) for Dyspnea
  * Description: Breathlessness severity measured by VAS.
  * Time Frame: Up to 15 days post-operative.
  * Unit of Measure: Units on a scale (0-10 cm).
  * Scale: 0 = no breathlessness, 10 = worst breathlessness imaginable; higher scores indicate worse dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Aziza M Mohammed, Head nurse, Study Chair — Woman's Health Hospital, Assiut University, Egypt
Locations (1):
- Woman's Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No